CLINICAL TRIAL: NCT02420262
Title: A Clinical Trial Comparing Efficacy and Safety of Insulin Degludec/Liraglutide (IDegLira) Versus Basal-bolus Therapy in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-4185; 2014-003621-18 (EudraCT Number); U1111-1160-6923 (Other: WHO); REec-2015-1682 (Registry Identifier: Spanish registry)
Record Dates: First submitted 2015-04-08; First posted 2015-04-17 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegLira (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- IGlar plus IAsp (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Once daily injected s.c./subcutaneously (under the skin) in combination with metformin.
  Arms: IDegLira
Drug: insulin glargine — Once daily injected s.c./subcutaneously (under the skin) in combination with metformin.
  Arms: IGlar plus IAsp
Drug: insulin aspart — Injected s.c./subcutaneously (under the skin) before each main meal.
  Arms: IGlar plus IAsp

SUMMARY:
This trial is conducted globally. The aim of this trial is to compare efficacy and safety of insulin degludec/liraglutide (IDegLira) versus basal-bolus therapy in combination with metformin in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing informed consent
* Type 2 diabetes subjects (diagnosed clinically) at least 6 months prior to screening
* HbA1c (glycosylated haemoglobin) 7.0-10.0% [53mmol/mol-86mmol/mol] (both inclusive) by central laboratory analysis
* Current treatment with IGlar (insulin glargine) for at least 90 calendar days prior to screening
* Stable daily dose of IGlar between 20 units and 50 units (both inclusive) for at least 56 calendar days prior to screening. Individual fluctuations of plus/minus 10% within the 56 calendar days prior to screening are acceptable, however on the day of screening total daily dose should be within the range of 20 units-50 units both inclusive
* Stable daily dose of metformin (at least 1500 mg or max tolerated dose) for at least 90 calendar days prior to screening
* Body mass index (BMI) below or equal to 40 kg/m^2

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 calendar days before screening
* Anticipated initiation or change in concomitant medications in excess of 14 calendar days known to affect weight or glucose metabolism, such as weight loss/modifying (e.g.; sibutramine, orlistat, thyroid hormones, corticosteroids)
* Impaired liver function, defined as alanine aminotransferase (ALT) at least 2.5 times upper limit of normal
* Renal impairment eGFR (electronic case report form) below 60 mL/min/1.73 m^2 as per CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration)
* Screening calcitonin at least 50 ng/L
* History of pancreatitis (acute or chronic)
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2015-07-26 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (105):
- United States (47):
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Bermuda Dunes, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Lincoln, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Natchitoches, Louisiana
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Jackson Heights, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Shelby, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Midlothian, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
- Argentina (4):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Salta
- Czechia (6):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Olomouc, Lazce
  - Novo Nordisk Investigational Site, Pardubice
  - Novo Nordisk Investigational Site, Prostějov
- France (11):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Bourgoin
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Coudray
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Saint-Priest-en-Jarez
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Vénissieux
- Greece (5):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Chalkida, Evia
  - Novo Nordisk Investigational Site, Ioannina
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (5):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Szombathely
  - Novo Nordisk Investigational Site, Tatabánya
- Israel (6):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Nahariya
  - Novo Nordisk Investigational Site, Rehovot
- Mexico (4):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Aguascalientes
  - Novo Nordisk Investigational Site, Durango
- Russia (4):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Volgograd
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bardejov
  - Novo Nordisk Investigational Site, Dolný Kubín
  - Novo Nordisk Investigational Site, Malacky
  - Novo Nordisk Investigational Site, Poprad
  - Novo Nordisk Investigational Site, Rožňava
- Spain (5):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Fuenlabrada - Madrid
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- [Result] Billings LK, Doshi A, Gouet D, Oviedo A, Rodbard HW, Tentolouris N, Gron R, Halladin N, Jodar E. Efficacy and Safety of IDegLira Versus Basal-Bolus Insulin Therapy in Patients With Type 2 Diabetes Uncontrolled on Metformin and Basal Insulin: The DUAL VII Randomized Clinical Trial. Diabetes Care. 2018 May;41(5):1009-1016. doi: 10.2337/dc17-1114. Epub 2018 Feb 26. PMID 29483185
- [Derived] Billings LK, Agner BFR, Altuntas Y, Gron R, Halladin N, Klonoff DC, Tentolouris N, Jodar E. The Benefit of Insulin Degludec/Liraglutide (IDegLira) Compared With Basal-Bolus Insulin Therapy is Consistent Across Participant Subgroups With Type 2 Diabetes in the DUAL VII Randomized Trial. J Diabetes Sci Technol. 2021 May;15(3):636-645. doi: 10.1177/1932296820906888. Epub 2020 Feb 28. PMID 32107930
- [Derived] Meneghini L, Doshi A, Gouet D, Vilsboll T, Begtrup K, Orsy P, Ranthe MF, Lingvay I. Insulin degludec/liraglutide (IDegLira) maintains glycaemic control and improves clinical outcomes, regardless of pre-trial insulin dose, in people with type 2 diabetes that is uncontrolled on basal insulin. Diabet Med. 2020 Feb;37(2):267-276. doi: 10.1111/dme.14178. Epub 2019 Nov 28. PMID 31705547
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 89 sites in 12 countries: Argentina (3 sites), Czech Republic (5 sites), France (3 sites), Greece (6 sites), Hungary (3 sites), Israel (6 sites), Mexico (3 sites), Russia (7 sites), Slovakia (5 sites), Spain (6 sites), Turkey (5 sites) and United States (37 sites).
Pre-assignment Details: Subjects with type 2 diabetes mellitus were on treatment with stable daily dose of insulin glargine (IGlar) between 20 units and 50 units (both inclusive) for at least 56 days prior to screening in combination with a stable daily dose of metformin (≥1500 mg or maximum tolerated dose) for at least 90 days prior to screening.
Groups:
- IDegLira: Insulin Degludec/Liraglutide (IDegLira: 100 U/3.6 mg per mL) was injected subcutaneously once daily (OD) for a duration of 26 weeks. IDegLira was supplied in a 3 mL pre-filled PDS290 pen-injector with a fixed IDeg/liraglutide ratio of 100 units/3.6 mg per mL solution. IDegLira treatment was initiated at 16 dose steps (containing 16 units IDeg /0.6 mg liraglutide) and adjusted twice weekly based on the mean of three pre-breakfast self-measured plasma glucose (SMPG) values measured on the days of the titration and the two days prior to the titration (target SMPG: 4.0-5.0 mmol/L [72- 90 mg/dL]).The maximum daily dose was 50 dose steps (50U IDeg /1.8 mg Lira). All subjects continued with metformin at pre-trial doses (≥ 1500 mg or the maximum tolerated dose), unless there was a safety concern.
- IGlar + IAsp: Subjects received insulin glargine plus prandial insulin aspart subcutaneously for duration of 26 weeks. A stable pre- trial OD dose of IGlar (20-50 units, in a 3 mL pre-filled Solostar®) was continued with metformin therapy (≥ 1500 mg or the maximum tolerated dose). IAsp was added to the IGlar therapy with a start dose of 4U using a 3 mL pre-filled FlexPen®, as prandial insulin treatment before each main meal. The dose of IGlar was adjusted twice weekly based on the mean of three pre-breakfast SMPG values measured on the days of the titration and the two days prior to the titration (target SMPG: 4.0-5.0 mmol/L [72- 90 mg/dL]). The dose of IAsp was titrated twice weekly based on pre-prandial and bedtime SMPGs, obtained on the three previous days (target SMPG: 4.0 - 6.0 mmol/L).
Period: Overall Study
Arm/Group | IDegLira | IGlar + IAsp
Started | 252 | 254
Exposed | 252 | 253 (One subject withdrew consent before exposure to trial product due to personal reasons.)
Completed | 250 | 249
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Unclassified | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects. The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised"
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegLira | IGlar + IAsp | Total
Number analyzed (Participants) | 252 | 254 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.0) | 58.0 (8.6) | 58.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 137 | 279
  Male | 110 | 117 | 227
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.21 (0.76) | 8.24 (0.81) | 8.22 (0.78)
Body Weight [Mean (Standard Deviation); unit: kg] | 87.2 (16.0) | 88.2 (17.2) | 87.7 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Change in HbA1c values after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". 8 subjects in IDegLira and 9 subjects in IGlar + IAsp arm did not contribute to the analysis for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated haemoglobin
Arm/Group | IDegLira | IGlar + IAsp
Number analyzed (Participants) | 244 | 245
Percentage of glycosylated haemoglobin | -1.48 (0.05) | -1.46 (0.05)
Statistical Analysis 1: Comparison: IDegLira vs IGlar + IAsp; Change from baseline in HbA1c was analysed using a mixed model for repeated measurements with an unstructured covariance matrix. The model included treatment, visit and region as fixed factors and baseline HbA1c as covariate. Interactions between visit and all factors and the covariate were also included in the model; Test type: Non-Inferiority or Equivalence — Non-inferiority for IDegLira vs basal-bolus (IGlar + IAsp) was considered confirmed if the upper boundary of the two-sided 95% confidence interval was strictly below 0.30% or equivalent for non-inferiority using one-sided test for null hypothesis (H0): D ≥0.30% against alternative hypothesis (HA): D <0.30% was less than or equal to 2.5%, where D is the mean treatment difference (IDegLira minus basal-bolus); p < 0.0001, Mixed Models Analysis; Treatment contrast = -0.02, 95% CI 2-sided [-0.16 to 0.12]

2. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemic Episodes.
Description: Severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe and/or BG confirmed by a plasma glucose value of <56 mg/dL (3.1 mmol/L), with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-26
Population: The safety analysis set (SAS) included all subjects receiving at least one dose of the investigational product or comparator. Subjects in the safety set contributed to the evaluation "as treated". One subject in IGlar + IAsp arm did not contribute to the analysis for this endpoint.
Measure: Number; unit: Number of episodes
Arm/Group | IDegLira | IGlar + IAsp
Number analyzed (Participants) | 252 | 253
Number of episodes | 129 | 975
Statistical Analysis 1: Comparison: IDegLira vs IGlar + IAsp; Hypoglycaemic episodes were analysed using a negative binomial regression. The model included treatment and region as fixed factors and logarithm of the time period in which a hypoglycaemic episode considered treatment emergent as offset. The test for superiority of the confirmatory secondary endpoints was carried out only if non-inferiority of IDegLira vs basal-bolus for primary endpoint was confirmed; Test type: Superiority or Other; p < 0.0001, Negative binomial regression model; Treatment ratio = 0.11, 95% CI 2-sided [0.08 to 0.17] — Superiority for IDegLira vs basal-bolus was considered confirmed if the 95% confidence interval for the treatment rate ratio was entirely below 1.0

3. Secondary Outcome: Change in Body Weight
Description: Change in body weight after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". 08 subjects in both IDegLira and IGlar + IAsp arm did not contribute to the analysis for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | IDegLira | IGlar + IAsp
Number analyzed (Participants) | 244 | 246
kg | -0.93 (0.22) | 2.64 (0.22)
Statistical Analysis 1: Comparison: IDegLira vs IGlar + IAsp; Body weight measurements were analysed using a linear mixed model with an unstructured covariance matrix. The model included treatment, visit and region as fixed factors and baseline bodyweight as covariate. Interactions between visit and all factors and the covariate were also included in the model. The test for superiority of the confirmatory secondary endpoints was carried out only if non-inferiority of IDegLira vs basal-bolus for primary endpoint was confirmed; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -3.57, 95% CI 2-sided [-4.19 to -2.95] — Superiority for IDegLira vs basal-bolus was considered confirmed if the 95% confidence interval for the treatment difference was below 0 or equal to zero

4. Secondary Outcome: Responder for HbA1c Below 7.0%
Description: Number of subjects with HbA1c below 7% after 26 weeks of treatment.
Time Frame: After 26 weeks of treatment
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". 14 subjects in IDegLira and 21 subjects in IGlar + IAsp arm did not contribute to the analysis for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegLira | IGlar + IAsp
Number analyzed (Participants) | 238 | 233
Participants
  Yes | 157 | 156
  No | 81 | 77

5. Secondary Outcome: Responder for HbA1c Below or Equal to 6.5 %
Description: Number of subjects with HbA1c below 6.5% after 26 weeks of treatment.
Time Frame: After 26 weeks of treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IDegLira | IGlar + IAsp
Number analyzed (Participants) | 238 | 233
Participants
  Yes | 118 | 104
  No | 120 | 129

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment (26 weeks + 7 days of follow-up).
Description: The safety analysis set (SAS) included all subjects receiving at least one dose of the investigational product or comparator. Subjects in the safety set contributed to the evaluation "as treated".
Arm/Group | IDegLira | IGlar + IAsp
Serious Adverse Events (participants affected / at risk) | 12/252 | 10/253
Other Adverse Events (participants affected / at risk) | 84/252 | 79/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=252) | IGlar + IAsp (N=253)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=252) | IGlar + IAsp (N=253)
Diabetic retinopathy (Eye disorders) | 9 (9) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 16 (24) | 10 (17)
Headache (Nervous system disorders) | 14 (17) | 18 (23)
Influenza (Infections and infestations) | 18 (21) | 12 (13)
Nasopharyngitis (Infections and infestations) | 12 (12) | 30 (35)
Nausea (Gastrointestinal disorders) | 28 (37) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.